CLINICAL TRIAL: NCT01860014
Title: Comparison of Two Different Natural Surfactants in the Treatment of Pulmonary Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Sami Ulus Children's Hospital (Other)
Responsible Party: Principal Investigator, Dilek Dilli, MD, Dr. Sami Ulus Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 306/29 March 2010; 306/29 March 2010 (Other: Ethics Committee)
Record Dates: First submitted 2013-05-20; First posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Pulmonary Hemorrhage
Keywords: Pulmonary hemorrhage; Mortality; Newborn
MeSH Terms: interventions — poractant alfa; beractant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beractant (Active Comparator): Beractant (Survanta): 100 mg/kg-intratracheal, just after pulmonary hemorrhage
  Interventions: Drug: Poractant alfa
- Poractant alfa (Active Comparator): Poractant alfa (Curosurf): 100 mg/kg-intratracheal, just after pulmonary hemorrhage
  Interventions: Drug: Beractant

INTERVENTIONS:
Drug: Poractant alfa — Curosurf: 100 mg/kg-intratracheal, just after pulmonary hemorrhage
  Other Names: Curosurf
  Arms: Beractant
Drug: Beractant — Survanta: 100 mg/kg-intratracheal, just after pulmonary hemorrhage
  Other Names: Survanta
  Arms: Poractant alfa

SUMMARY:
The incidence of pulmonary hemorrhage (PH) was about 1.3 per 1,000 live births. PH occurs mainly in preterm ventilated infants with severe respiratory distress syndrome (RDS) who often have a PDA and have received surfactant. Although not clear, the cause of PH is thought to be due to a rapid lowering of intrapulmonary pressure, which facilitates left to right shunting across a patent ductus arteriosus and an increase in pulmonary blood flow. Prospective uncontrolled studies that used surfactant for PH in neonates have shown promising results in treating PH.In this study we aimed to evaluate the effect of two different natural surfactants in neonates with pulmonary hemorrhage.

DETAILED DESCRIPTION:
The incidence of PH was about 1.3 per 1,000 live births. Formerly,the risk factors associated with PH included the severity of the associated illness, intrauterine growth restriction, patent ductus arteriosus (PDA), coagulopathy, and the need for assisted ventilation. Currently, PH occurs mainly in preterm ventilated infants with severe respiratory distress syndrome (RDS) who often have a PDA and have received surfactant. Currently, PH complicates the hospital course of 3-5% of preterm infants with RDS. The cause of PH is thought to be due to a rapid lowering of intrapulmonary pressure, which facilitates left to right shunting across a patent ductus arteriosus and an increase in pulmonary blood flow. Prospective uncontrolled studies that used surfactant for PH in neonates have shown promising results in treating PH.In this study we aimed to evaluate the effect of two different natural surfactants in neonates with pulmonary hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants <1500 g
* Within first week of life

Exclusion Criteria:

* Major congenital abnormalities
* Without parental consent

Ages: 1 Hour to 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Oxygen requirement | 6 hour
  We will evaluate the need of oxygen support within 6 hour after surfactant

SECONDARY OUTCOMES:
Mortality | 4 weeks
  We will compare the rate of mortality between the groups during neonatal period

CONTACTS AND LOCATIONS:
Overall Officials: Şenol Bozdağ, MD, Principal Investigator — Zekai Tahir Burak Hospital
Locations (1):
- Zekai Tahir Burak Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Rogers D. Pulmonary haemorrhage, surfactant, and low-birthweight babies. Lancet. 1993 Mar 13;341(8846):698. doi: 10.1016/0140-6736(93)90469-w. No abstract available. PMID 8095608